CLINICAL TRIAL: NCT07343297
Title: Ask Questions About Clinical Trials (ASQ - CT): An Implementation Trial of a Communication Intervention to Improve Patient-Provider Communication About Clinical Trials and Provider Invitations to Clinical Trials
Brief Title: Ask Questions About Clinical Trials
Acronym: ASQ-CT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Lauren Hamel, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-082
Record Dates: First submitted 2025-12-15; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Oncology; Cardiac Disease; Neurologic Disorder
MeSH Terms: conditions — Neoplasms; Heart Diseases; Nervous System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ask Questions about Clinical Trials (ASQ-CT) Brochure (Experimental): Ask Questions about Clinical Trials (ASQ-CT), a clinical trial communication intervention brochure
  Interventions: Behavioral: Ask Questions about Clinical Trials brochure

INTERVENTIONS:
Behavioral: Ask Questions about Clinical Trials brochure — Communication intervention called a question prompt list

SUMMARY:
The overall goal of this study is to assess the implementation of the Ask Questions about Clinical Trials (ASQ-CT) brochure, a patient-focused communication tool previously demonstrated to improve patient-provider communication about clinical trials. Participants will be given the ASQ-CT brochure at Time 1 (baseline) and participants will complete a questionnaire at three timepoints, baseline (Time 1), Pre-Research Visit (Time 2), and Post-Research Visit (Time 3).

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal to 18 years
* Appointment to see a provider at a Karmanos Cancer Institute-McLaren or a medical encounter at McLaren Center for Research and Innovation (MCRI) site for medical/systemic treatment
* Potentially eligible for a clinical trial
* Speak and read English well enough to be able to understand consent documents and complete surveys

Exclusion Criteria:

* Not able to complete study documents on their own physically or cognitively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-05 (Estimated)

PRIMARY OUTCOMES:
Effectiveness - Self-Efficacy in managing patient-provider interactions - Quantitative Scale | From Baseline (Time 1) to end of Pre-Clinic Visit (Time 2)
  Improvement of self-efficacy in managing patient-providers interactions between baseline (Time 1) and pre-clinic visit (Time 2). Measured using scale of 1-5 where a higher score is equal to a better outcome

SECONDARY OUTCOMES:
Reach - Number and Proportion | At start of Participation
  Proportion of individuals invited to participate who agree to participate. The denominator will be the absolute number of individuals who are identified and approached as potential participants; the numerator will be the number of people who agreed to participate. Investigators will track the number of people who were excluded from participation and why. Investigators anticipate that reach will vary by research site and patient baseline characteristic (i.e., sociodemographic, health literacy level). These variations between clinics will be based only on consented participants. Although the Investigators will track refusals, data will not be collected from patients who decline.
Effectiveness - Self-Efficacy in managing patient-provider interactions - Quantitative Scale | From Pre-Clinic (Time 2) to end of Post-Clinic Visit (Time 3) up to 3 months.
  Improvement of self-efficacy in managing patient-providers interactions between baseline (Time 2) and pre-clinic visit (Time 3). Measured using scale of 1-5 where a higher score is equal to a better outcome
Effectiveness - Knowledge - Quantitative Scale | From Baseline (Time 1) to end of Pre-Clinic Visit (Time 2)
  Improvement of knowledge between baseline (Time 1) and pre-clinic visit (Time 2). Measured using scale of 1-5 where a higher score is equal to a better outcome.
Effectiveness - Knowledge - Quantitative Scale | From Pre-Clinic Visit (Time 2) to end of Post-Clinic Visit (Time 3) up to 3 months
  Improvement of knowledge between pre-clinic visit (Time 2) and post-clinic visit (Time 3). Measured using scale of 1-5 where a higher score is equal to a better outcome
Effectiveness - Trust - Quantitative Scale | From Baseline (Time 1) to end of Pre-Clinic Visit (Time 2)
  Improvement in trust in providers between baseline (Time 1) and pre-clinic visit (Time 2). Measured using scale of 1-5 where a higher score is equal to a better outcome
Effectiveness - Trust - Quantitative Scale | From Pre-Clinic Visit (Time 2) to end of Post-Clinic Visit (Time 3) up to 3 months
  Improvement in trust in providers between pre-clinic visit (Time 2) and post-clinic visit (Time 3). Measured using scale of 1-5 where a higher score is equal to a better outcome
Effectiveness - distress - Quantitative Scale | From Baseline (Time 1) to end of Pre-Clinic Visit (Time 2)
  Improvement in distress between baseline (Time 1) and pre-clinic visit (Time 2). Measured using scale of 1-5 where a higher score is equal to a worse outcome.
Effectiveness - distress - Quantitative Scale | From Pre-Clinic Visit (Time 2) to end of Post-Clinic Visit (Time 3) up to 3 months
  Improvement in distress between pre-clinic visit (Time 2) and post-clinic visit (Time 3). Measured using scale of 1-5 where a higher score is equal to a worse outcome.
Adoption - Number and Proportion | At start of Participation
  Adoption is defined by the number, proportion, and representativeness of the clinics willing to implement the Ask Questions about Clinical Trials (ASQ-CT) brochure. The denominator will be the absolute number of clinics who are invited to implement the ASQ-CT brochure; the numerator will be the number of clinics who agree to implement the ASQ-CT brochure.
Implementation of the Intervention | From Baseline (Time 1) to up to 3 months
  Implementation is defined as intervention agents' (e.g., research/clinic staff) fidelity to the adaptations of the intervention and associated implementation strategies. Patients will receive the Ask Questions about Clinical Trials (ASQ-CT) brochure in Time 1. In Time 2, patients will be asked to respond to two fidelity (yes/no) questions, including: 1. When the participant received the ASQ-CT brochure, did the participant receive instructions on how to use it from the clinic/research staff (yes/no)? Was the participant given the chance to discuss the ASQ-CT brochure with clinic/research staff (yes/no?)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Hamel, PhD, MBA, Principal Investigator — Wayne State University